CLINICAL TRIAL: NCT06357390
Title: Physiologic and Clinical Effect of High-flow Oxygen Therapy in Tracheostomized Patients With Prolonged Mechanical Ventilation Undergoing Weaning Trials
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202106174RINB
Record Dates: First submitted 2021-12-29; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-07

CONDITIONS: High Flow Oxygen Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is aimed at patients who have been admitted to the respiratory care center of this hospital who meet the PMV conditions (defined as continuous use of the ventilator for at least ten days) who are about to receive the ventilator out of training. After obtaining the explanatory consent, they will undergo continuous complete Before and after spontaneous breathing training, collect various relevant physiological data of lung volume and ventilation perfusion distribution, and analyze and predict the correlation of ventilator detachment.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 20 years old, have undergone tracheotomy, have been using a ventilator for at least 10 days, and have stable vital signs.

Exclusion Criteria:

* Age <20 years
* The oxygen concentration (FiO2) provided by the respirator exceeds 60%
* pregnant
* Blood pressure-systolic blood pressure below 70 mmHg
* Heartbeat is lower than 50/min or higher than 160/min
* Respiration rate is higher than 50/min
* Lack of voluntary breathing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were transferred to RCC and tried to get out of the ventilator after tracheotomy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
ventilation perfusion distribution measurement | 16 weeks
  1. Within 2 hours before starting the whole day of ATC, start measuring lung volume and ventilation perfusion distribution in SIMV+PS mode.
  2. Start the 72-hour ATC mode, measure once within 2 hours; measure again after 24 hours.
  3. Within 2 hours before and after the completion of the 72-hour ATC conversion to the 24-hour tracheostomy tube high flow oxygen, one measurement is made.
  4. Measure once within 2 hours before and after the completion of 24-hour high-flow oxygen conversion to 5 consecutive days of spontaneous breathing training.
  5. After the use of high flow oxygen starts, measure it every 24 hours until the 5th day.

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Shuin Jerng, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan